CLINICAL TRIAL: NCT05105711
Title: Evaluating the Feasibility of a Mobile Coaching Intervention to Improve HPV Vaccine Delivery
Brief Title: Mobile Coaching to Improve HPV Vaccine Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Kaiser Permanente (Other); University of Minnesota (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-0810; 1R21CA241518-01 (NIH)
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: HPV Vaccine; Provider Communication Practices; Vaccine Recommendation Practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary care providers (Experimental): Providers who treat 11-12 year old adolescent patients in participating Kaiser Permanente Washington pediatric and family medicine practices.
  Interventions: Behavioral: QI coaching intervention

INTERVENTIONS:
Behavioral: QI coaching intervention — The intervention consists of two main components: a webinar communication workshop and use of the Checkup Coach mobile app. The Checkup Coach intervention begins with a brief (<1 hour), communication training workshop that reviews evidence on HPV vaccination, models guideline-consistent recommendations, trains providers to address parent concerns, and facilitates discussion of shared goals for improving. Next, providers are invited to download and use the Checkup coach mobile app at their discretion for the 12-week study period. Providers complete in-app self-assessments and receive tailored feedback about their HPV vaccine recommendation quality, progress toward improving recommendation practices, a dashboard of aggregate HPV vaccination coverage for patients in their clinic, and tips for addressing parents' concerns about HPV vaccination every time they use the app.

SUMMARY:
The purpose of this study is to examine the feasibility of using Checkup Coach, a mobile coaching intervention, to improve the way that primary care providers recommend HPV vaccination to adolescent patients and their parents. To conduct this feasibility study, the investigators will deliver the Checkup Coach intervention to 20 Kaiser Permanente Washington primary care providers who routinely recommend HPV vaccine to adolescent patients. The investigators will use a single-arm, pre-post design. Participating primary care providers will attend a 1-hour virtual communication workshop and then use a mobile phone app to receive additional coaching for 12 weeks. Providers will complete surveys at three time points: before the communication workshop, immediately after the workshop, and at 12-week follow-up. Surveys will assess changes in providers' self-reported HPV vaccine recommendation practices and beliefs about HPV vaccine and also acceptability of the intervention. The investigators hypothesizes that providers' HPV vaccine communication will improve between baseline and 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Primary care providers who treat 11-12 year old adolescent patients in participating Kaiser Permanente Washington pediatric and family medicine practices

Exclusion Criteria:

* Primary care providers who do not treat adolescent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Gilkey, PhD, Principal Investigator — University of North Carolina
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Providers who treat adolescent patients in participating Kaiser Permanente Washington primary care clinics in the Puget Sound and Spokane region. 21 participants consented, with 19 completing the study and 2 not completing the study.
Pre-assignment Details: Providers were eligible and worked in clinics that agreed to participate in the study.
Period: Overall Study
Arm/Group | Primary Care Providers
Started | 21
Completed | 19
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Primary Care Providers
Number analyzed (Participants) | 19
Age, Customized [Count of Participants; unit: Participants]
  >18 years | 19
  <18 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 4
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 19
Mean recommendation quality score [Mean (Full Range); unit: units on a scale] — Providers' mean composite score on a 5-item index of self-reported use of HPV vaccine communication practices with scores ranging from 5-25 (5 indicating the lowest quality score to 25 indicating the highest quality score). Population: Only participants who completed all parts of the intervention and follow-up were included in analyses
  units on a scale | 23.4 [18 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Change in HPV Vaccine Recommendation Quality Score
Description: The change in providers' mean composite score on a 5-item index of self-reported use of HPV vaccine communication practices with scores ranging from 5-25 (5 indicating the lowest quality score to 25 indicating the highest quality score).
Time Frame: Baseline, 12 weeks
Population: Primary care providers who participated in the Checkup Coach QI workshop and who completed data collection at all three time points
Measure: Mean (Full Range); unit: score
Arm/Group | Primary Care Providers
Number analyzed (Participants) | 19
score
  Baseline | 23.4 [18 to 25]
  Follow-up | 24.2 [17 to 25]

ADVERSE EVENTS:
Description: Adverse even data was not collected because it was a one time educational training and mobile phone educational intervention to use at participants' discretion. This was for a quality improvement project and did not pose any risk to participants.
Groups:
- Experimental: Primary Care Providers: Providers who treat 11-12 year old adolescent patients in participating Kaiser Permanente Washington pediatric and family medicine practices. Adverse events were not collected.
Arm/Group | Experimental: Primary Care Providers
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT05105711/Prot_SAP_000.pdf